CLINICAL TRIAL: NCT00439855
Title: Enoxaparin Versus Unfractionated Heparin in PCI
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Triemli Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZEUS
Record Dates: First submitted 2007-02-23; First posted 2007-02-26 (Estimated); Last update posted 2007-02-26 (Estimated); Status verified 2007-02

CONDITIONS: Coronary Artery Disease
Keywords: Enoxaparin, heparin, hemorrhages
MeSH Terms: conditions — Coronary Artery Disease; Hemorrhage | interventions — Heparin

INTERVENTIONS:
Drug: Enoxaparin i.v.
Drug: unfractionated heparin

SUMMARY:
Enoxaparin 0.75mg/kg BW is not inferior to weight adjusted unfractionated heparin as anticoagulation for PCI

ELIGIBILITY:
Inclusion Criteria:

* PCI for stable ischemia or ACS

Exclusion Criteria:

* Cardiogenic shock,
* Pretreatment with study drugs,
* Lack of informed consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2100
Dates: Start 2003-09; Study Completion 2006-02

PRIMARY OUTCOMES:
Quadruple endpoint: death, MI, urgent TVR, major bleeding

SECONDARY OUTCOMES:
major bleeding, minor bleeding, thrombocytopenia

CONTACTS AND LOCATIONS:
Overall Officials: osmund bertel, MD, Principal Investigator — Division of Cardiology Triemli Hospital Zurich
Locations (1):
- Division of Cardiology Triemli Hospital Zurich, Zurich, Switzerland